CLINICAL TRIAL: NCT05059132
Title: Tele-rehabilitation Following Curative Intent Therapy of Lung Cancer
Brief Title: Inspiratory Muscle Training and Behavioral Support to Alleviate Dyspnea and Promote Walking in Lung Cancer Survivors: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCD-820773
Record Dates: First submitted 2021-09-13; First posted 2021-09-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lung Neoplasm
Keywords: Pilot study; Tele-rehabilitation; Remote rehabilitation; Exercise therapy; Aerobic exercise; Physical activity
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: This is a pilot, parallel randomized study of an exercise + behavioral support intervention to reduce dyspnea and improve walking behavior among lung cancer survivors following curative intent therapy. Forty participants will be randomized 1:1 to the intervention or control arm, with assessments of feasibility, acceptability, safety, and patient-centered outcomes. The intervention period is 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation (Experimental): Participants in the tele-rehabilitation arm will receive a home-based, remotely delivered rehabilitation program.
  Interventions: Behavioral: Tele-rehabilitation
- Education only (Active Comparator): Participants in the education arm will receive educational materials only, delivered through telecommunication messages.
  Interventions: Other: Education only

INTERVENTIONS:
Behavioral: Tele-rehabilitation — The tele-rehabilitation intervention will include education, inspiratory muscle training, and behavioral support to promote walking.
  Arms: Tele-rehabilitation
Other: Education only — The education only arm will receive information on the importance of general exercise following lung cancer treatment.
  Arms: Education only

SUMMARY:
This is a pilot randomized study to investigate the feasibility, acceptability, safety, and effects of a novel tele-rehabilitation intervention for stage I-IIIA lung cancer survivors following curative intent therapy.

The specific aims and hypotheses are:

Specific Aim 1: Conduct a pilot, phase IIb, parallel randomized (1:1) study to investigate the feasibility, acceptability, and safety of inspiratory muscle training and behavioral support to promote walking in tele-rehabilitation with stage I-IIIA lung cancer survivors following curative intent therapy (N=40).

Hypothesis 1a: ≥ 20% eligible patients will enroll; ≥75% of participants will achieve ≥75% adherence to the tele-rehabilitation program.

Hypothesis 1b: ≥75% of participants will perceive tele-rehabilitation as acceptable (Telemedicine Satisfaction and Usefulness Questionnaire ≥4). There will be 0 intervention adverse events.

Specific Aim 2: Explore the effects of the tele-rehabilitation program (N=40).

Hypothesis 2: At 12 weeks, participants in the tele-rehabilitation (experimental) arm, compared to education only (control) arm, will have a trend of greater improvements in outcomes, including:

1. accelerometry-measured physical activity (primary outcome); and
2. functional capacity, self-reported physical activity, control of dyspnea and anxiety symptoms, sleep quality, and quality of life (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* history of stage I-IIIA lung cancer;
* completed curative intent therapy (i.e., lung cancer resection surgery, definitive radiation, or concurrent chemoradiation) within 1-6 months;
* access to a mobile phone or personal computer with internet access;
* willingness to wear activity trackers

Exclusion Criteria:

* dementia (or cognitive impairment identified by chart review) resulting in inability to follow directions or provide written informed consent;
* acute myocardial infarction, ventricular tachycardia, ventricular fibrillation, acute cerebrovascular event, or acute asthma exacerbation in past 2 months;
* spontaneous pneumothorax in past 12 months;
* Parkinson's disease;
* multiple sclerosis;
* amyotrophic lateral sclerosis;
* additional movement/gait disorders that may be identified by chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in change in accelerometry-measured physical activity between baseline and week 12 | Baseline, mid study (week 6), and end of study (week 12).
  Physical activity will be measured by the activPAL4 device (PAL Technologies, Ltd).

SECONDARY OUTCOMES:
Difference in change in functional capacity between baseline and week 12 | Baseline, mid study (week 6), and end of study (week 12)
  Functional capacity will be measured using the mobile six-minute walk test.
Difference in change in self-reported physical activity between baseline and week 12 | Baseline, mid study (week 6), and end of study (week 12)
  Self-reported physical activity will be measured using the International Physical Activity Questionnaire - Short Form
Difference in change in control of dyspnea between baseline and week 12 | Baseline, mid study (week 6), and end of study (week 12)
  Dyspnea control will be measured using the the University of California, San Diego Shortness of Breath Questionnaire.
Difference in change in anxiety symptoms between baseline and week 12 | Baseline, mid study (week 6), and end of study (week 12)
  Anxiety symptoms will be measured using the General Anxiety Disorder-7
Difference in change in sleep quality between baseline and week 12 | Baseline, mid study (week 6), and end of study (week 12)
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index
Difference in change in quality of life between baseline and week 12 | Baseline, mid study (week 6), and end of study (week 12)
  Quality of life will be measured using the St. George's Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ha DM, Comer A, Dollar B, Bedoy R, Ford M, Gozansky WS, Zeng C, Arch JJ, Leach HJ, Malhotra A, Prochazka AV, Keith RL, Boxer RS. Telemedicine-based inspiratory muscle training and walking promotion with lung cancer survivors following curative intent therapy: a parallel-group pilot randomized trial. Support Care Cancer. 2023 Sep 1;31(9):546. doi: 10.1007/s00520-023-07999-7. PMID 37656252